CLINICAL TRIAL: NCT05718778
Title: Single-arm, Open, Exploratory Clinical Study on the Safety and Efficacy of Piamprilimab (AK105) Combined With Radiotherapy for Neoadjuvant Treatment of Soft Tissue Sarcoma
Brief Title: Piamprilizumab (AK105) Combined With Radiotherapy for Neoadjuvant Treatment of Soft Tissue Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Associate chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLXFZ-001
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Piamprilizumab (AK105) combined with radiotherapy for neoadjuvant treatment of soft tissue sarcoma (Experimental): Piamprilizumab (AK105) combined with radiotherapy for neoadjuvant treatment of soft tissue sarcoma
  Interventions: Drug: Piamprimab (AK105)

INTERVENTIONS:
Drug: Piamprimab (AK105) — Piamprilizumab (AK105) combined with radiotherapy for neoadjuvant treatment of soft tissue sarcoma
  Other Names: radiotherapy

SUMMARY:
The primary objective of this study was to evaluate the safety and efficacy of paamprilimab combined with radiotherapy for neoadjuvant treatment of soft tissue sarcoma. The primary endpoint was pathological complete response rate (CPR).

DETAILED DESCRIPTION:
31 patients with stage I, II, and III resectable soft tissue sarcoma were enrolled in this study at the Bone and soft Tissue Ward 1 of Henan Cancer Hospital. The main objective of this study was to evaluate the safety and efficacy of paamprimab combined with radiotherapy for neoadjuvant treatment of soft tissue sarcoma. The primary endpoint of this study was pathological complete response rate (CPR).

ELIGIBILITY:
Inclusion Criteria:

1. Age :18-70 years old, gender unlimited;
2. Histopathologically confirmed patients with stage I, II, and III resectable soft tissue sarcomas (subtypes These include undifferentiated pleomorphic sarcoma, angiosarcoma, fibrosarcoma, synovial sarcoma, and smooth muscle Sarcoma);
3. No previous treatment with radiotherapy, chemotherapy, antiangiogenic drugs or immune checkpoint inhibitors To cure;
4. Measurable lesions at baseline according to Recist version 1.1:
5. ECOGPS:0-2, expected survival greater than 6 months.
6. If the major organs are functioning normally, the following criteria are met:

   Hemoglobin (Hb)≥ 90g/L, neutrophil (ANC)≥1.5×109/L, Platelet count (PLT)≥ 80×109/L, Serum creatinine (Cr)≤ 1.5× upper limit of normal (ULN) or creatinine clearance (CCr)≥60ml/min; Total bilirubin (TB)≤ 1.5ULN; Aminotransferase (AST) and alanine aminotransferase (ALT)≤ 2.5×ULN; Left ventricular ejection fraction ≥50%;
7. Women of childbearing age must have been using reliable contraception or have had a pregnancy test (serum or urine) with negative results within 7 days prior to inclusion and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last test drug administration. For men, consent was required to use an appropriate method of contraception or to have been surgically sterilized during the trial period and within 8 weeks after the last administration of the trial drug
8. Sign an informed consent form (or legal representative sign) to demonstrate that they understand the purpose of the study and the procedures required by the Institute, and are willing to participate in the study.

Exclusion Criteria:

1. Previous chemoradiotherapy, use of antiangiogenic drugs or other immune checkpoint inhibitors;
2. Have any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy).
3. Patients with vitiligo or childhood asthma that has been completely resolved and can be admitted as adults without any intervention; Patients requiring medical intervention with bronchodilators are not included;
4. Patients with congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active B (HBVDNA≥500IU/mL), hepatitis C (HCV antibody positive, and HCV-RNA higher than the detection limit of analysis method) or co-infection of hepatitis B and hepatitis C;
5. Use of immunosuppressive drugs within 14 days prior to initial use of the study drug, excluding intranasal and inhaled corticosteroids or systemic steroid stimulants at physiological doses (i.e., not exceeding 10mg/ day prednisone or its equivalent);
6. Live attenuated vaccine administered within 4 weeks prior to initial administration or planned for the study period;
7. Other malignant tumors in the past 3 years;
8. Imaging (CT or MRI) showed the presence of tumors invading local great vessels, or accompanied by the formation of tumor thrombus in great veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava);
9. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy;
10. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal medical treatment); Patients with newly diagnosed angina pectoris or myocardial infarction within 3 months prior to screening; Arrhythmias (including QTcF: male ≥450ms, female ≥470ms) requiring long-term use of antiarrhythmic drugs and New York Heart Association grade ≥II cardiac insufficiency;
11. Severe cardiovascular disease, such as New York Heart Society Heart disease (Grade II or higher), myocardial infarction, cerebrovascular accident, unstable arrhythmia, unstable angina in the 3 months prior to enrollment, Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria, or left ventricular ejection fraction <50%, must be treated with a stable treatment regimen as best determined by the treating physician, with consultation with a cardiologist if necessary;
12. A severe infection occurring within 4 weeks prior to initial administration (e.g., requiring intravenous antibiotic, antifungal, or antiviral medication), or an unexplained fever >38.5°C during screening/prior to initial administration;
13. A history of idiopathic pulmonary fibrosis, institutional pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia on chest CT scan at screening;
14. Had gastrointestinal or non-gastrointestinal fistula before enrollment (≥ grade 3);
15. Known history of allogeneic organ transplantation or allohematopoietic stem cell transplantation;
16. Pregnant or lactating women; Fertile patients are unwilling or unable to use effective contraception A doer;
17. Known allergic reaction, hypersensitivity or intolerance to test drugs and their excipients;
18. Subjects who are participating in another clinical study or whose first drug use is less than 4 weeks after the end of the previous clinical study (final drug use), or who have 5 half-lives of the investigational drug;
19. Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders;
20. Any condition that the investigator considers to be prejudicial to the subject or to the subject's inability to meet or perform the study requirements exists.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | From the start of treatment to surgery at week 12
  From the beginning of treatment to the completion of surgery

SECONDARY OUTCOMES:
Progression-free survival | It takes about 12 weeks from the start of treatment to surgery
  From the start of treatment to the progression of the disease
Overall survival | 0 to 120 months
  From the beginning of treatment to death

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No